CLINICAL TRIAL: NCT06509932
Title: Feasibility Study of Jefcare Sterile Medical Sheets for the Prevention of Incontinence-associated Dermatitis and the Maintenance of Local Skin Microclimate Stability in Adult Patients in the Intensive Care Unit
Brief Title: Prevention of Incontinence-associated Dermatitis and Maintenance of Local Skin Microclimate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20240161
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-07

CONDITIONS: Incontinence-associated Dermatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jefcare Sterile Medical Sheets (Experimental): Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: Jefcare Sterile Medical Sheets and skin care regimen.
  Interventions: Device: Jefcare Sterile Medical Sheets
- Molicare Premium Bed Mat (Other): Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: MoliCare Premium Bed Mats and skin care regimen.
  Interventions: Device: MoliCare Premium Bed Mats

INTERVENTIONS:
Device: Jefcare Sterile Medical Sheets — Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: Jefcare Sterile Medical Sheets and skin care regimen.
  Arms: Jefcare Sterile Medical Sheets
Device: MoliCare Premium Bed Mats — Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: MoliCare Premium Bed Mats and skin care regimen.
  Arms: Molicare Premium Bed Mat

SUMMARY:
To explore the feasibility of Jefcare Sterile Medical Sheets in preventing incontinence-associated dermatitis and maintaining a stable local skin microclimate in adult patients in the intensive care unit.

DETAILED DESCRIPTION:
Jefcare Sterile Medical Sheet is an incontinence care product designed by researchers following the Expert consensus on the clinical application of disposable absorbent care products for adults with incontinence. The product has good laboratory test indicators and has the potential to prevent incontinence-associated dermatitis and maintain the stability of the local skin microclimate. Still, there is a lack of high-quality clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Intensive care unit incontinent patients (incontinence time ≥2 days)
2. Age ≥18 years
3. patients at high risk of IAD (Perineal Assessment Tool ≥ 7)
4. Voluntarily participate in the study and sign an informed consent form. If the subject is unable to read and sign the informed consent form due to incapacitation or other reasons, their guardian is required to represent the informed process and sign the informed consent form. If the subject is unable to read the informed consent form (e.g., illiterate subjects), a witness will be required to witness the informed process and sign the informed consent form.

Exclusion Criteria:

1. Patients who have developed IAD
2. Expected subsequent stay in the intensive care unit <5 days
3. Use of nappies, pull-ups, incontinence pads, etc.
4. Simple urinary incontinence with indwelling catheterization, external urinary bag without leakage; simple fecal incontinence with built-in drainage device, external ostomy bag, OB tampon without leakage; double incontinence with indwelling catheterization, external urinary bag, built-in drainage device, external ostomy bag, OB tampon without leakage.
5. The IAD may affect the skin area within the scope of the disease that affects the IAD judgment.
6. The IAD may affect the skin area within the scope of the skin breaks, infection
7. Patients who are not suitable for turning and cannot tolerate the side-lying position.
8. Patients with known allergies or keloid scarring
9. Women who are known to be pregnant or breastfeeding or who are planning to have a baby during the study period.
10. Patients who have participated in a clinical trial of another drug or medical device within 3 months.
11. Patients who, in the opinion of the investigator, are not suitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of IAD | Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  incidence of IAD = number of cases of patients with IAD in the group/total number of patients in the group × 100%.

SECONDARY OUTCOMES:
The time of IAD occurrence | Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  Time to IAD after enrolment
The site and severity of IAD occurrence | Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  IAD may affect a range of 14 skin regions. A patient was considered to have IAD onset as long as the patient had IAD in 1 place.
  Using the IAD categorization tool, the tool classifies the severity of IAD into 3 levels. level 0 is represented by intact skin, no redness, and no difference in comparison to the skin of other body parts. level 1 is represented by red, intact, and possibly erythematous skin with edema. level 2 is represented by red, broken, and possibly skin with edema, blisters, blisters, vesicles, eruption of the skin, excoriation, and infected skin.
The skin microclimate and skin barrier function | Total 2 times. 1 prior to intervention, 1 on occurrence of IAD or end of the study i.e. day 5 of the intervention.
  Examination site: the lower abdomen/pubic arch; the inner right thigh; the inner left thigh ; the lower left buttock; the lower right buttock.
  Examination indicators: Skin temperature , skin hydration, skin PH , melanin , erythema , transepidermal water loss. Three measurements were taken at each site and averaged.
Date of faecal incontinence (ICU admission to end of study);Mean number of faecal incontinence per day (ICU admission to end of study);The average number of medical sheets used per day. | The average number of medical sheets used per day:Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  Date of faecal incontinence (ICU admission to end of study) = total number of days of fecal incontinence after ICU admission.
  Date of faecal incontinence (ICU admission to end of study) = Total number of fecal incontinence episodes after ICU admission/total number of days of fecal incontinence after ICU admission.
  Average number of medical sheets used per day = total number of medical sheets used/time of intervention.
Mycological examination | Total 2 times. 1 prior to intervention, 1 on occurrence of IAD or end of study i.e. day 5 of the intervention.
  A cotton swab impregnated with saline sampling solution was applied to the local skin in a circular pattern from the upper left buttock, gluteal cleft, upper right buttock, lower right buttock, posterior right thigh, posterior left thigh, lower left buttock, and perineum in a sequential order, and the sampling cotton swabs were rotated accordingly, and the swabs were applied to the plate after sampling. Then to the front of the patient, a cotton swab was taken in a circular pattern from the lower abdomen/pubic arch, the left inguinal fold between the genitals and the thighs, the left inner thigh, the right inner thigh, the right inguinal fold between the genitals and the right thigh, and the genitals in the order of applying a localized skin and the subsequent rotation of the sampling cotton swab, and the swabs were applied to the plate after sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyang Hu, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China